CLINICAL TRIAL: NCT04448301
Title: PC001 - Study to Evaluate the Usability of PointCheck, a Novel Optical Technology for Screening Non-Invasively Severe Neutropenia
Brief Title: PC001- A Study to Evaluate the Usability of PointCheck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leuko Labs, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-39964
Record Dates: First submitted 2020-06-11; First posted 2020-06-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms; Neutropenia
Keywords: Medical Device; Technology; Non-invasive
MeSH Terms: conditions — Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PointCheck Cohort (Experimental)
  Interventions: Diagnostic Test: PointCheck

INTERVENTIONS:
Diagnostic Test: PointCheck — This is a usability study on PointCheck, a new technology to detect chemotherapy-induced neutropenia

SUMMARY:
This a study about the usability of PointCheck a novel non-invasive technology for monitoring chemotherapy-induced neutropenia.

The study will include patients with cancer visiting the outpatient hematology clinic for their standard of care chemotherapy administration. A final sample size of 90 oncologic outpatients will be enrolled and studied with the technology.

The main objective is to evaluate the usability of PointCheck. Secondary outcomes include a preliminary assessment of PointCheck diagnostic accuracy and precision.

For this, study subjects will be tested twice with PointCheck during the same session and the usability in an at-home simulated environment by naïve users will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study and to provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
2. Male or Female aged 18 years or above.
3. Diagnosed with a hematological (e.g., lymphoma, myeloma) or breast cancer.
4. Scheduled active treatment with cytotoxic chemotherapy with an associated high/intermediate risk of neutropenia.
5. Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria

1. Participants with amputations, congenital malformations, or any severe abnormalities of the hands as determined by the investigator.
2. Participants with a history of vasculitis, Raynaud syndrome, scleroderma, mixed connective tissue disease or any other rheumatologic systemic condition that could produce microcirculatory changes in the nailfold.
3. Participants with circulating tumour cells in previous or current lab determinations.
4. Participants with leukemia.
5. Participants with any condition producing significant tremor (e.g., essential tremor, Parkinson´s disease, dystonic tremor).
6. Inadequately medically controlled hypotension (systolic blood pressure <90 and diastolic blood pressure < 60mmHg).
7. Participants whose gold standard blood differential was obtained more than 120 minutes after the last evaluation with the medical device.
8. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
9. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
PointCheck's Usability | Up to two-weeks
  To gather data with the ultimate goal of determining the usability of the proposed non-invasive method measured by the number of errors of correct videos acquired for analyses.
System Usability Scale (0-100 higher scores indicates better usability) | Up to three-weeks
  To confirm the usability of the system using the System Usability Scale

SECONDARY OUTCOMES:
PointCheck's Precision | Up to two-weeks
  To perform an exploratory analysis of the precision of PointCheck's estimation of neutropenia status from two independent one-minute videos.
PointCheck's Accuracy | Up to three-weeks
  To perform a exploratory analysis of PointCheck's accuracy (e.g., sensitivity, specificity, predictive values) to detect severe neutropenia compared with the gold standard blood analysis method employed by Boston Medical Center core laboratory in the range between ≤500 and >500 absolute neutrophil count/µL.
PointCheck's Utility | Up to three-weeks
  To evaluate the number of patients that had to be rescheduled because the sole presence of neutropenia and how many of them were correctly detected with PointCheck.
Number of participants with device-related adverse events as assessed by CTCAE v5.0 | Up to three-weeks
  To confirm PointCheck's safety determining the % of AEs and SAEs related to the device use.

OTHER OUTCOMES:
Diagnostic performance for a second cutoff | Up to three-weeks
  The preliminary diagnostic accuracy to detect grade III neutropenia according to CTCAE V5 (<1000 ANC/mm3) measured by the sensitivity and the specificity will be the evaluated with reference to the corresponding laboratory measures acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sloan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamaj G, Pablo-Trinidad A, Butterworth I, Bell N, Benasutti R, Bourquard A, Sanchez-Ferro A, Castro-Gonzalez C, Jimenez-Ubieto A, Baumann T, Rodriguez-Izquierdo A, Pottier E, Shelton A, Martinez-Lopez J, Sloan JM. Usability Evaluation of a Noninvasive Neutropenia Screening Device (PointCheck) for Patients Undergoing Cancer Chemotherapy: Mixed Methods Observational Study. J Med Internet Res. 2022 Aug 9;24(8):e37368. doi: 10.2196/37368. PMID 35943786